CLINICAL TRIAL: NCT02402517
Title: Pulse EnRiched Food and Exercise Clinical Trials (PERFECT Project): Part 2 - Acute Effects of Pulse Ingredients in Food Products on Aerobic Endurance and Substrate Oxidation During Exercise, as Well as, the Blood Glucose, Insulin, Lactate and Food Intake Response Following an Endurance Exercise Session in Adults - Study 1
Brief Title: PERFECT Project - Part 2 - Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Saskatchewan Pulse Growers (Other); Alberta Pulse Growers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: B2014:114-2
Record Dates: First submitted 2014-12-17; First posted 2015-03-30 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2017-05

CONDITIONS: Diabetes; Obesity
Keywords: Diabetes Prevention; Obesity Prevention
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Extruded snack control (Placebo Comparator): 100% corn flour
  Interventions: Other: Control
- Extruded snack with small particle size pea flour (Experimental): 60% corn flour and 40% small particle size pea flour
  Interventions: Other: Small particle size pea flour
- Extruded snack with large particle size pea flour (Experimental): 60% corn flour and 40% large particle size pea flour
  Interventions: Other: Large particle size pea flour
- Extruded snack with lentil flour (Experimental): 60% corn flour and 40% lentil flour
  Interventions: Other: Lentil flour
- Extruded snack navy bean flour (Experimental): 60% corn flour and 40% navy bean flour
  Interventions: Other: Navy bean flour
- Extruded snack with pinto bean flour (Experimental): 60% corn flour and 40% pinto bean flour
  Interventions: Other: Pinto bean flour

INTERVENTIONS:
Other: Control — Non pulse extruded snack
  Arms: Extruded snack control
Other: Small particle size pea flour — Pulse extruded snack
  Arms: Extruded snack with small particle size pea flour
Other: Large particle size pea flour — Pulse extruded snack
  Arms: Extruded snack with large particle size pea flour
Other: Lentil flour — Pulse extruded snack
  Arms: Extruded snack with lentil flour
Other: Navy bean flour — Pulse extruded snack
  Arms: Extruded snack navy bean flour
Other: Pinto bean flour — Pulse extruded snack
  Arms: Extruded snack with pinto bean flour

SUMMARY:
The objectives are to test the acute effects of different extruded pulse snacks on: 1) aerobic endurance and substrate oxidation during exercise 2) response of blood glucose, insulin and appetite on an aerobic exercise session, and 3) food intake two hours following the exercise session. The investigators hypothesize that consumption of food products containing pulse ingredients 60 minutes before exercise will increase aerobic endurance (lower oxygen consumption), decrease carbohydrate oxidation (greater respiratory quotient), and a reduction in lactate production during compared to the same exercise session following the ingestion of a non-pulse food. The investigators also hypothesize that consumption of extruded pulse snacks will lead to lower blood glucose, insulin, appetite and food intake, suggesting lower calorie compensation, following a 60-minute aerobic exercise session compared to the same exercise session following the ingestion of a non-pulse food.

ELIGIBILITY:
Inclusion Criteria:

* Normoglycemic (<5.6 mmol/L) and normotensive (systolic blood pressure <140 mm Hg and diastolic blood pressure below < 90 mm Hg)
* BMI of 18.5-29.9 kg/m2

Exclusion Criteria:

* Restrained eaters
* Regularly skip breakfast
* Smokers
* Those who are active (organized activities or athletic training at a high intensity; ≥ 150 min per week of moderate to vigorous physical activity)
* Those on medications that may influence study outcomes or have experienced any gastrointestinal related health conditions/surgeries over the past year.
* Those unable to walk for an hour continuously

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose and Insulin Concentrations | 0 - 240 min
  Measured in blood using intravenous catheter at 14 time points, used to calculate area under curve (AUC). Glucose will be determined by automated methods using Abbot Spectrum CCX Analyzer, and Insulin will be measured by commercially available RIA kits. (Composite measure)
Food Intake | at 120 min
  Ad-libitum meal. Food consumed measured by weight.
Subjective Appetite | 0-240 min
  Measured by VAS questionnaire at 14 time points, used to calculate area under curve (AUC).( Composite measure)
Exercise intensity | 60 minutes
  Sixty minute exercise protocol at minutes 60 to 120. Oxygen consumption measured during exercise at 3 time points.

SECONDARY OUTCOMES:
Lactate concentration | 60 minutes
  60 minute exercise protocol at minutes 60 to 120. Measured before, during, and exercise exercise at 3 time points
Palatability of treatments | at 5 minutes
  Measured by VAS questionnaire
Palatability of meal | at 260 minutes
  Measured by VAS questionnaire
Physical comfort | 0-240 min
  Measured by VAS questionnaire at 13 time points, used to calculate area under curve (AUC) (Composite measure)
Energy/fatigue | 0-240 min
  Measured by VAS questionnaire at 13 time points, used to calculate area under curve (AUC) (Composite measure)
Heart rate | 60-120 min
  Heart rate monitored over a 60 minute exercise protocol. To monitor exercise intensity and give a measure of fatigue (cardiovascular drift)
Substrate Oxidation | 60 minutes
  Measured during 60 minute exercise protocol at minutes 60-120. Respiratory quotient measured during exercise at 3 time points.

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PhD, Principal Investigator — University of Manitoba, Richardson Centre for Functional Foods and Nutraceuticals
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada